CLINICAL TRIAL: NCT01949363
Title: The Pharmacokinetics of Extended Duration High-Dose Cefixime for the Decreased Susceptibility of Neisseria Gonorrhoeae: A Phase I Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-0025; HHSN272201500007I
Record Dates: First submitted 2013-09-19; First posted 2013-09-24 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2015-06

CONDITIONS: Gonorrhoea
Keywords: Gonococcal Infections, Cefixime, Neisseria gonorrhoeae, Azithromycin, antibiotic, cephalosporin
MeSH Terms: conditions — Gonorrhea | interventions — Cefixime

ARMS (2):
- Stage 2 (Cohorts C and D) (Experimental): Cohort C will first be given 1200mg cefixime orally once; Cohort D will be given 800mg cefixime orally three times (every 8 hours); 6 subjects in each cohort
  Interventions: Drug: Cefixime
- Stage 1 (Cohorts A and B) (Experimental): Cohort A will be given 400mg of cefixime orally once; Cohort B will be given 800mg of cefixime given orally once; 6 subjects in each cohort
  Interventions: Drug: Cefixime

INTERVENTIONS:
Drug: Cefixime — Cefixime is an FDA approved oral semi-synthetic cephalosporin antibiotic. The standard dose (400mg), high dose (800mg and 1200mg), and multiple 800mg and 1200mg doses given over a 24-hour period using a dose-frequency escalation method. Cohort A receives 400 mg orally once, Cohort B receives 800 mg orally once; Cohort C receives 1200 mg orally once; Cohort D receives 800 mg orally 3 times (every 8 hrs)

SUMMARY:
This study is a Phase I, open label, non-randomized, dose-frequency escalation pharmacokinetics study among 24 healthy male and female subjects, aged 18 to 45 years to determine the pharmacokinetics and safety of high-, multi-dose cefixime for the treatment of reduced susceptibility gonorrhea. Stage 1(Cohorts A and B) will examine the pharmacokinetics of single 400mg and 800mg dose of cefixime. Stage 2(Cohorts C and D) subjects will take 800mg of cefixime every 12 hours for 2 doses. If that dosing regimen is well tolerated, the dose-frequency will escalate to 800mg every 8 hours for 3 doses, and serum levels of cefixime will be measured. Study duration is approximately 47 weeks.

DETAILED DESCRIPTION:
This study is a Phase I, open label, non-randomized, dose-frequency escalation pharmacokinetics study among 24 healthy male and female subjects, aged 18 to 45 years to determine the pharmacokinetics and safety of high multi-dose cefixime for the treatment of reduced susceptibility gonorrhea. The study will occur in two stages as described below. Stage 1: Confirm/establish the pharmacokinetics (PK) of 400mg and 800mg doses of cefixime tablet. Stage 2: Define dosing frequency necessary to achieve total serum cefixime levels that exceed 2.0 mcg/mL for over 20 hours. Stage 1 (Cohorts A and B): Six subjects will be admitted to the Johns Hopkins Bayview Clinic Trials Unit to assess each dosing regimen, for a total of 12 subjects. At time=0, subjects will undergo baseline serum cefixime levels, followed by ingestion of cefixime. Serum collections will occur at times 0, 1, 2, 4, 8, 12, 16, 20, and 24 hours. Cohort B will have the same serum collection time points as Cohort A. Cohorts A & B will be run nearly simultaneously as logistically feasible. Stage 2 (Cohorts C and D): After determining the PK parameters of single dose 800mg, the PK simulation model will be repeated, adjusting the model as needed based on findings from study Stage 1. Assuming there are no major discrepancies between Figure 2 (above) and the new PK simulations, the following regimens will be tested, beginning with Cohort C. Six subjects per dosing regimen, Cohorts C and D, will be admitted to the Johns Hopkins Bayview Medical Center, for a total of 12 subjects. The 800mg q12 hour x 2 regimen (Cohort C) will be tested first. For Cohort C, serum cefixime levels will be drawn at 12, 16, and 26 hours. If the q12 regimen is deemed safe and tolerable after review by the SMC, Cohort D will commence with the 800mg q8 hour x 3 regimen. Total serum cefixime levels will be drawn for Cohort D at 8, 16, 20 and 26 hours (see Section 7.2). All Stages, All Cohorts: All samples collected for PK analysis will be shipped to the University of Toledo, Dr. Jeffrey Blumer's HPLC lab for processing. Specimens will be analyzed by high performance liquid chromatography (HPLC) for total cefixime concentration levels. Targeted clinical evaluations will be used to monitor for subject reported side effects. Subjects will be asked about specific symptoms they may have experienced, including abdominal pain, nausea, vomiting, diarrhea, flatulence, headache, and rash, or any other symptoms. Additionally, subjects will be asked to maintain a Subject Diary (Appendix E) from Study Day 0 through Day 7 to record information about any symptoms experienced or medications taken. Study duration is approximately 47 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects between 18 and 45 years, inclusive
* Ability to understand the consent process and procedures
* Informed consent obtained and signed
* Body mass index (BMI) < 35 kg/m^2
* Subjects agree to be available for all study visits
* Negative Breathalyzer
* Agreement by female subjects with reproductive potential to use an adequate method of contraception during the study and for 30 days after study drug administration. Female subjects must agree to the use of TWO reliable methods of contraception while receiving study drug and for 30 days after study drug administration if sexually active, which can include: condoms, spermicidal gel, diaphragm, hormonal or non-hormonal intrauterine device, surgical sterilization, oral contraceptive pill (OCP), and depot progesterone injections.

Exclusion Criteria:

* Subjects who take any prescription medication on a regular basis (except oral contraceptives, OCPs), including but not limited to, anti-psychotics, anti-depressants, anti-epileptics, cardiac medications, anti-hypertensives etc.
* Medical condition that precludes participation, including the following:
* Hypertension with confirmed systolic blood pressure >140 mmHg or confirmed diastolic blood pressure >90 mmHg, measured after 10 - 15 minutes of rest
* Morbid obesity (BMI>/=35)
* Current diagnosis of pulmonary disease
* History of or current diagnosis of diabetes
* Autoimmune disorder, such as lupus, Wegener's, rheumatoid arthritis
* History of malignancy except low-grade skin cancer, (i.e., basal cell carcinoma thought to be cured)
* Known diagnosis of prolonged QT interval
* History of alcohol abuse
* History of seizure disorder
* History of renal disease
* Chronic renal, hepatic, or pulmonary disease or other condition that could interfere with the absorption of the study drug or predispose to adverse gastrointestinal events (e.g., surgical resection of significant proportions of the stomach or bowel, gastric bypass, gastric banding, irritable bowel syndrome, inflammatory bowel disease)
* Positive serology results for HIV, HBsAg, or HCV antibodies
* Subjects who have taken any prescription drugs in the previous 14 days or within 5 half-lives before dosing
* Ingestion of over the counter medications or herbal supplements within 7 days of dosing
* Positive urine toxicology for marijuana, cocaine, amphetamines, opiates, PCP, barbiturates or benzodiazepines
* History of allergic reaction or intolerance to cephalosporins
* History of allergic reaction to penicillin (all stages)
* Subjects with an allergy to macrolides may not participate in Stage 3
* Subjects with QTc >450ms (Fridericia's correction) on screening ECG may not participate in Stage 3.
* Positive pregnancy test; pregnant or nursing women
* Screening laboratory tests outside of the acceptable limits presented in Appendix C
* Any specific condition that, in the judgment of the Investigator, precludes participation because it could affect subject safety

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2013-12; Primary Completion 2015-02 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Total serum concentrations of cefixime at multiple time points for both individuals and cohorts in total | Day 1, 2 and Day 7
Safety and tolerability assessed by laboratory monitoring, targeted clinical evaluations,: serum chemistries, liver functions tests (LFTs), hematology panel, coagulation panel, and urinalysis | Screening to Day 7
Pharmacokinetic curves of cefixime levels versus time: time to peak drug level, half-life, and elimination rate | Day 0-1, 2 and Day 7
Pharmacokinetic curves of cefixime levels versus time: total time that cefixime levels exceed 4x the MIC of 0.5 mcg/mL(serum level of 2.0 mcg/mL) | Day 0-1, 2 and Day 7
Pharmacokinetic curves of cefixime levels versus time: total area under the curve (AUC) | Day 0-1, 2 and Day 7
Pharmacokinetic curves of cefixime levels versus time: peak cefixime level. | Day 0-1, 2 and Day 7
Pharyngeal fluid concentrations of cefixime for Cohorts C - D: Cmax and ratio of fluid to serum concentration | Day 0-1
Assess subject reported adverse events, unsolicited symptoms and discomforts | Up to Day 30

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Bayview Medical Center - Infectious Diseases, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Barbee LA, Nayak SU, Blumer JL, O'Riordan MA, Gray W, Zenilman JM, Golden MR, Griffiss JM. A Phase 1 Pharmacokinetic and Safety Study of Extended-Duration, High-dose Cefixime for Cephalosporin-resistant Neisseria gonorrhoeae in the Pharynx. Sex Transm Dis. 2018 Oct;45(10):677-683. doi: 10.1097/OLQ.0000000000000844. PMID 29624558